CLINICAL TRIAL: NCT01412931
Title: Protein and Ultrasound Indicators of Preterm Birth
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0570
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervicovaginal fluid and placental membranes will be retained for study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1) Pregnant women with a single intrauterine pregnancy: 50 women with uncomplicated pregnancies and no history of preterm birth.
- 2) Pregnant women with a single intrauterine pregnancy: 50 multiparous women with history of spontaneous preterm labor or preterm premature rupture of membranes (PPROM).
- 3) Pregnant women with a single intrauterine pregnancy: 20 women evaluated on the labor and delivery unit because they are deemed to be at high risk for preterm birth.

SUMMARY:
Women are being asked to participate in a research study that is looking for new methods to understand and predict premature birth (birth before 37 weeks of pregnancy-full term pregnancy is 40 weeks). In this study the investigators will be looking at proteins in vaginal fluid, tissue from the placenta after the baby is born (fetal membranes), and a new form of ultrasound of the mouth of the womb (cervix) that measures its length, volume, and stiffness, in order to try to know who will have a preterm birth and who will reach full term. The investigators will collect the vaginal fluid samples and perform ultrasounds both in the clinic throughout pregnancy in normal women, and from women admitted to the hospital because they are in early labor. The investigators will collect the placental tissue after the baby is born (this is normally discarded). This study will help us to understand the process of preterm birth and the investigators hope that this will eventually allow us to develop better methods to treat preterm labor and prevent the birth of premature babies.

ELIGIBILITY:
Inclusion Criteria:

* Single live intrauterine pregnancy
* Good gestational age dating

Exclusion Criteria:

* History of prior cervical procedure such as LEEP, CKC, or cryotherapy
* Maternal or fetal indication for preterm delivery
* Cerclage in place

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women with a single intrauterine pregnancy with good gestational age dating, and live fetus with no indications for preterm delivery will be enrolled. Three groups of subjects will be recruited: a) 50 women with uncomplicated pregnancies and no history of preterm birth, b) 50 multiparous women with history of spontaneous preterm labor or preterm premature rupture of membranes (PPROM) c) 20 women evaluated on the labor and delivery unit because they are deemed to be at high risk for preterm birth. Pregnant women of all races and ethnicities will be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in Serial Elastography Measurements | Groups a and b, ultrasound imaging and CVF collection will occur no more than four times with one week spacing between assessments. Group "d" will be assessed more frequently (up to 1× per day).
  Serial elastography measurements will enable us to quantify changes in tissue modulus and structure longitudinally through normal, term pregnancy.

SECONDARY OUTCOMES:
Changes in Biomechanical and biochemical analyses of the chorioamnion | Groups a and b, ultrasound imaging and CVF collection will occur no more than four times with one week spacing between assessments. Group "d" will be assessed more frequently (up to 1× per day).
  To quantify the strength and related mechanical properties, characterize the composition of the extracellular matrix, and characterize the secreted protein profile.
Correlation of Protein and biochemical analysis of the cervicovaginal fluid (CVF) | Groups a and b, ultrasound imaging and CVF collection will occur no more than four times with one week spacing between assessments. Group "d" will be assessed more frequently (up to 1× per day).
  Protein and biochemical analysis of the CVF, and correlation with cervical tissue stiffness and morphology, will enable detection of specific bio-markers that are present during normal and premature cervical ripening.
Stratification of Ultrasound parameters, chorioamnion biomechanical and biochemical properties, and CVF proteins . | Groups a and b, ultrasound imaging and CVF collection will occur no more than four times with one week spacing between assessments. Group "d" will be assessed more frequently (up to 1× per day).
  Identify specific values and biomarkers able to identify patients at risk of preterm labor and preterm birth.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Ferguson, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States